CLINICAL TRIAL: NCT01363674
Title: Easypod Connect: A National, Multicentre, Observational Registry to Study Adherence and Long Term Outcomes of Therapy in Paediatric Subjects Using Easypod™ Electromechanical Device for Growth Hormone Treatment in Greece
Brief Title: To Assess the Level of Adherence of Subjects Receiving SAIZEN® Via Easypod™ in Greece
Acronym: ECOS GRE
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck A.E., Greece (Industry)
Responsible Party: Sponsor
Other Study IDs: EMR 200104-520
Record Dates: First submitted 2011-05-30; First posted 2011-06-01 (Estimated); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Growth Disorders
Keywords: Growth disorders; Saizen; Easypod; Growth hormone; Pediatric subject
MeSH Terms: conditions — Growth Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Easypod™ — Saizen (Somatotropin) as per Summary of Product Characteristics administered by Easypod™
  Other Names: Saizen; Somatotropin

SUMMARY:
This is a National, Multicentre, Observational Registry to study adherence and long term outcomes of therapy in paediatric subjects using Easypod™ electromechanical device for growth hormone treatment from hospitals in Greece and to assess the level of adherence of subjects receiving SAIZEN® via Easypod™.

DETAILED DESCRIPTION:
Subjects will be enrolled in a multicenter, longitudinal observational registry. Parents/subjects will provide their Informed Consent/assent to upload their data for populationbased analyses and optionally to adhere to a patient adherence support program designed to improve their adherence and, ultimately, clinical outcomes. Adherence data will be primarily derived from the Easypod™ device combined with physician data entry of outcome measures. Data will be collected retrospectively and prospectively. This will allow the establishment of adherence profiles and explore the hypothesis that patient adherence support programs improve adherence and subsequent clinical outcomes. Collected data will be also analyzed in a multinational pooled analysis of comparable national studies.

Primary Objective:

- To assess the level of adherence of subjects receiving SAIZEN® via Easypod™

Secondary Objectives:

* To identify adherence subject profiling
* To describe the impact of adherence on clinical outcomes for subject receiving SAIZEN® via Easypod™
* To asses the impact of adherence on Insulin-like Growth Factor 1 (IGF1) (i.e. above, below or within normal ranges)
* To assess/describe the impact of the Greek Scientific Service (Patient Support Program)

ELIGIBILITY:
Inclusion Criteria:

* Administered growth hormone (SAIZEN®) via the Easypod™ auto-injector, according to approved Summary of Product Characteristics (SmPC)
* Naïve subjects or already treated with SAIZEN® and Easypod™ for up to 1 year
* Male and female between 2 - 18 years of age, or over 18 without fusion of growth plates
* Parent's or guardian's (or subject's if over 18 without fusion of growth plates) written informed consent, given before entering data into the registry, with the understanding that the subject or parent/guardian may withdraw consent at any time without prejudice to future medical care.

Exclusion Criteria:

* Subjects taking growth hormone in whom growth plates have fused (i.e. for taking growth hormone for its metabolic effects)
* Contra-indications to SAIZEN® as defined in the approved SmPC
* Use of an investigational drug or participation in another interventional clinical study

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Paediatric subjects (aged 2-18) who are taking SAIZEN® for registered indications using the Easypod™ electromechanical device.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2013-04-30 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Mean percent of adherence by subject | At least 6 months and up to 5 years

SECONDARY OUTCOMES:
Correlation of adherence and growth outcome after each year of SAIZEN® treatment with Easypod™ | At least 6 months and up to 5 years
  Correlation of adherence and growth outcome (height velocity (HV), height velocity-standard deviation score (HV-SDS), height, change in height (height SDS) after each year of SAIZEN® treatment with Easypod™
Subject adherence profile based on age, gender, indication, self-injection or not, time on treatment | At least 6 months and up to 5 years
Correlation of adherence with current IGF-I status (i.e. above, below or within normal ranges) | At least 6 months and up to 5 years
Impact of Greek Scientific Service (Patient Support Program) on adherence and outcomes for subjects using Easypod™. | At least 6 months and up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck A.E., Greece
Locations (1):
- For Recruiting Locations in Greece,, Please Contact the Merck KGaA Communication Center, Greece

REFERENCES:
- [Result] Koledova, E. et al. (2017) Analysis of results from the global, 5-year Easypod™ Connect Observational Study (ECOS) study in children with growth disorders. 10th International Meeting for Pediatric Endocrinology; 2017 Sep 14-17; Washington, DC.
- [Result] Wit, JM. et al. (2017) Effect of adherence on the 2-year growth response to growth hormone treatment in prepubertal children with idiopathic isolated growth hormone deficiency participating in the EasypodTM Connect Observational Study (ECOS). 10th International Meeting of Paediatric Endocrinology; 2017 Sep 14-17; Washington, DC.
- [Derived] Charmandari E, Vlachopapadopoulou E, Kyritsi EM, Sakellariou D, Koledova E, Nespithal K, Michalacos S. Adherence and long-term outcomes of therapy in paediatric patients in Greece using the easypod electromechanical device for growth hormone treatment: The phase IV multicentre easypod connect observational study (ECOS). Growth Horm IGF Res. 2020 Aug-Oct;53-54:101336. doi: 10.1016/j.ghir.2020.101336. Epub 2020 Jul 18. PMID 32739654